CLINICAL TRIAL: NCT02542670
Title: Genetic Variants of Selected Genes Using Target Deep Sequencing in Colo-Rectal Cancer Patients.
Brief Title: Genetic Variants of Selected Genes in Colo-Rectal Cancer Patients.
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Sherief Abd-Elsalam (Other)
Collaborators: Tanta University (Other)
Responsible Party: Sponsor-Investigator, Sherief Abd-Elsalam, Lecturer, Tanta University
Organization: Tanta University (Other)
Other Study IDs: Dr Said Hammad
Record Dates: First submitted 2015-09-02; First posted 2015-09-07 (Estimated); Last update posted 2017-07-26 (Actual); Status verified 2017-07

CONDITIONS: Cancer Colon
MeSH Terms: conditions — Colonic Neoplasms | interventions — Whole Genome Sequencing

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Biospecimen Retention: Samples With DNA — At least 50 ng of tumor DNA will be extracted from FFPE samples and/or fresh tissue and used for hybridization capture and NGS using the IlluminaMiSeqDx platform.
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (3):
- Cancer colon with no distant metastasis: Genetic: Whole genome Sequencing
  Interventions: Genetic: Whole genome sequencing
- Cancer colon with distant metastases: Genetic: Whole genome Sequencing
  Interventions: Genetic: Whole genome sequencing
- control group: Genetic: Whole genome Sequencing
  Interventions: Genetic: Whole genome sequencing

INTERVENTIONS:
Genetic: Whole genome sequencing — At least 50 ng of tumor DNA will be extracted from FFPE samples and/or fresh tissue and used for hybridization capture and NGS using the IlluminaMiSeqDx platform.

SUMMARY:
Colorectal cancers (CRC) are the third most common human malignancy, and are also the leading cause of cancer related deaths worldwide. Early detection of premalignant lesions such as adenomatous polyps has decreased the risk of CRCs; however, cases which are initially undetected and progress to advanced CRC with distant metastasis are still unfortunately incurable. The development of CRC is a complex and heterogeneous process arising from an interaction between multiple etiological factors, including genetic factors and environmental factors such as diet and lifestyle. The challenges are to understand the molecular basis of individual susceptibility to colorectal cancer and to determine factors that initiate the development of the tumor, drive its progression, and determine its responsiveness or resistance to antitumor agents. Next generation sequencing(NGS)-driven genomic studies are already reporting novel features of cancer genomes beyond the traditional mutational categories. Recent advance in sequencing technology has enabled comprehensive profiling of genetic alterations in CRC.These methods are facilitating an increase in the efficiency and resolution of detection of each of the principal types of somatic cancer genome alterations, including nucleotide substitutions, small insertions and deletions, copy number alterations, chromosomal rearrangements,DNA methylation sequencing such as bisulfite-sequencing and microbial infections. Besides the microsatellite instability (MSI), some researchers reported novel mitochondrial mutations in the cancer genomes. NGS technology will help the investigators for understanding of entire CRC genomes and the obtained knowledge will lead to a better diagnosis and personalized targeted therapeutics for CRC management

DETAILED DESCRIPTION:
Identification of the problem:Colorectal cancers (CRC) are the third most common human malignancy, and are also the leading cause of cancer related deaths worldwide. Early detection of premalignant lesions such as adenomatous polyps has decreased the risk of CRCs; however, cases which are initially undetected and progress to advanced CRC with distant metastasis are still unfortunately incurable. The development of CRC is a complex and heterogeneous process arising from an interaction between multiple etiological factors, including genetic factors and environmental factors such as diet and lifestyle. The challenges are to understand the molecular basis of individual susceptibility to colorectal cancer and to determine factors that initiate the development of the tumor, drive its progression, and determine its responsiveness or resistance to antitumor agents. Next generation sequencing(NGS)-driven genomic studies are already reporting novel features of cancer genomes beyond the traditional mutational categories. Recent advance in sequencing technology has enabled comprehensive profiling of genetic alterations in CRC.These methods are facilitating an increase in the efficiency and resolution of detection of each of the principal types of somatic cancer genome alterations, including nucleotide substitutions, small insertions and deletions, copy number alterations, chromosomal rearrangements,DNA methylation sequencing such as bisulfite-sequencing and microbial infections. Besides the microsatellite instability (MSI), some researchers reported novel mitochondrial mutations in the cancer genomes.NGS technology will help the investigators for understanding of entire CRC genomes and the obtained knowledge will lead to a better diagnosis and personalized targeted therapeutics for CRC management.Experimental design: The study design to attempt to identify the unique mutational spectrum and novel targets of genomic, epigenetic alterations in Egyptian colorectal cancer patients in Delta Regionusing Whole Exome and Epigenetic deep sequencing.Expected results:NGS-based genome analysis facilitates the identification of unrecognized gene mutation of Egyptian CRC cancer especially in Delta Region which may be biologically different from Western CRC as the environmental factors are different.Significance of the expected results:The results of this project will benefit in(1) Identification of novel features or mutation types in CRC genomes In Delta Region. (2) Understanding the advancement of pathway-level in colorectal carcinogenesis and (3) Identify Clinically relevant genetic and epigenetic biomarkers for noninvasive diagnosis and clinically actionable targets for personalized targeted medicine.

ELIGIBILITY:
Inclusion Criteria:

1. Ages Eligible for Study: 10 Years and older
2. Genders Eligible for Study: Both
3. Patients who can give informed consent themselves
4. 10 healthy controls will also be included in the study.

Exclusion Criteria:

1. Other cancer types rather than CRC.
2. Younger age than 10 years

Min Age: 10 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Cancer colon with no distant metastasis Cancer colon with distant metastases control group
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2015-07 (Actual); Primary Completion 2019-12 (Estimated); Study Completion 2019-12 (Estimated)

PRIMARY OUTCOMES:
Number of cancer patients with abnormal genetic mutations . | 2 years
  Number of cancer patients having abnormal genetic mutations .

CONTACTS AND LOCATIONS:
Overall Officials: Said Hammad abdou, Prof, Principal Investigator — Prof of clincal pathology and genetics; Samah mosaad aboelenein, lecturer, Study Director — lecturer of gastroenterology and hepatology; Asem Elfert, Prof, Study Chair — Prof of gastroenterology and hepatology; Sherief Abd-Elsalam, Lecturer, Study Chair — lecturer of gastroenterology and hepatology; Walaa Elkhalawany, Lecturer, Study Chair — lecturer of gastroenterology and hepatology; Nehal Elmashad, Prof, Study Chair — Prof of oncology; Mohamed Labib Salem, Prof, Study Chair — Prof of immunology and genetics; Abdel-Aziz Zidan, lecturer, Study Chair — lecturer of immunology and genetics; Amira youssef, lecturer, Study Chair — Lecturer of clinical pathology; Ayman Elsaka, prof, Study Chair — Prof of pathology; Gamal Mousa, prof, Study Chair — Prof of general surgery; Khalil Abas, Prof, Study Chair — Prof of public health and medical statistics; Osama Elkhadrawy, Prof, Study Chair — Prof of general surgery; Eman Ebrahim Ebrahim Farghal, Ph.D., Study Chair — Tanta University; Marwa H Saied, Ph.D., Study Chair — Tanta University
Locations (2):
- Egypt (2):
  - Sherief Abd-Elsalam, Cairo
  - Tanta university hospital, Cairo

IPD SHARING:
Plan to Share IPD: Undecided